CLINICAL TRIAL: NCT03403543
Title: Chinese Pregnant Woman Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Liangkun Ma, Obstetrics and Gynecology, Peking Union Medical College Hospital
Other Study IDs: PUMC-CPWCS
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Pregnancy Related; Pregnancy Disease; Pregnancy; Infant; Risk Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: This cohort study only set up a group. We will follow up and observe the pregnant women's lifestyle during pregnancy in order to find the risk factors of adverse pregnancy outcomes. We will divide the participants into more than one group according to the variables（e.g. age, smoking status, drinking status, sleep pattern .etc.）

SUMMARY:
Purpose To determine the relationship between maternal lifestyle and obstetric and neonatal outcomes.

Methods and analysis This is a multicentre, prospective, cohort study including more than 5000 participants in 24 hospitals in 12 provinces from July 2017 to July 2018 in China. Maternal lifestyle (environmental exposures, diet, physical activity, sleeping, psychology and economics) and metabolic status will be collected by the electronic self-administered questionnaire at the first, second and third trimesters and 42 days postpartum, respectively. Obstetric and neonatal outcomes and metabolic status recorded by a clinical research coordinator. Descriptive statistics will be used to investigate the outcomes of maternal and newborn across China. Logistical regression and covariance analysis will be used to determine the relationship between maternal lifestyle and obstetric and neonatal outcomes. SAS statistical software will be used for data analysis.

Ethics and dissemination Permission for the study was obtained from Chinese Academy of Medical Sciences and Peking Union Medical College. Ethics approval was obtained from the Ethics Review Committee at Department of Scientific Research, Peking Union Medical College Hospital, Beijing, China. The results will be published in peer-reviewed journals or disseminated through conference presentations.

ELIGIBILITY:
The participants were pregnant women who satisfied the following criteria: (1) ≥16 years old; (2) at 5-12 weeks' gestational; (3) able to complete the questionnaire; (4) permanent residents in the study locations; and (5) willing to sign the consent form.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only pregnant women at 5-12weeks gestationnal will be included in this study
Study Population: More than 5000 pregnant women will be recruited from July 2017 to July 2018 during their routine antenatal check at the first trimester. Maternal lifestyle (environmental exposure, diet, nutrient, physical activity, sleep quality, psychology and economics) are collected by electronic self-administered questionnaire at the first, second, third and 42 days postpartum. A clinical research coordinator will record the metabolic status (pre-pregnancy BMI and GWG) and obstetric and neonatal outcomes will be recorded.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
preterm birth | 2017.10.1-2019.3.1
  The doctors will record the delivery time
birth weight | 2017.10.1-2019.3.1
  The doctors will record the birth weight
birth defects | 2017.10.1-2019.3.1
  The doctors will record the birth defects

CONTACTS AND LOCATIONS:
Overall Officials: Yu Jiang, doctor, Principal Investigator — School of Public Health, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun Y, Shen Z, Zhan Y, Wang Y, Ma S, Zhang S, Liu J, Wu S, Feng Y, Chen Y, Cai S, Shi Y, Ma L, Jiang Y. Investigation of optimal gestational weight gain based on the occurrence of adverse pregnancy outcomes for Chinese women: a prospective cohort study. Reprod Biol Endocrinol. 2021 Aug 30;19(1):130. doi: 10.1186/s12958-021-00797-y. PMID 34461936
- [Derived] Lyu T, Chen Y, Zhan Y, Shi Y, Yue H, Liu X, Meng Y, Jing A, Qu Y, Ma H, Huang P, Man D, Li X, Wu H, Zhao J, Shan G, Jiang Y. Cohort profile: the Chinese Pregnant Women Cohort Study and Offspring Follow-up (CPWCSaOF). BMJ Open. 2021 Mar 23;11(3):e044933. doi: 10.1136/bmjopen-2020-044933. PMID 33757952
- [Derived] Sun Y, Shen Z, Zhan Y, Wang Y, Ma S, Zhang S, Liu J, Wu S, Feng Y, Chen Y, Cai S, Shi Y, Ma L, Jiang Y. Effects of pre-pregnancy body mass index and gestational weight gain on maternal and infant complications. BMC Pregnancy Childbirth. 2020 Jul 6;20(1):390. doi: 10.1186/s12884-020-03071-y. PMID 32631269